CLINICAL TRIAL: NCT01675024
Title: A Single-site, Single-dose and Multiple-dose Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of Rotigotine Transdermal Patch in Healthy Chinese Subjects.
Brief Title: Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of Rotigotine Transdermal Patch in Healthy Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SP0913
Record Dates: First submitted 2012-08-27; First posted 2012-08-29 (Estimated); Last update posted 2012-12-04 (Estimated); Status verified 2012-12

CONDITIONS: Healthy
Keywords: Neupro, Pharmacokinetics, healthy Chinese subjects
MeSH Terms: interventions — rotigotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rotigotine, Period 1 (Experimental): In Period 1 (Day 1 to Day 3) all 24 subjects will receive only 1 dose 2 mg / 24 hours.
  Interventions: Drug: Rotigotine, Period 1
- Rotigotine, Period 2 (Experimental): In Period 2 (Day 7 to Day 14) all 24 subjects will receive 2 mg / 24 hours for 3 days then 4 mg / 24 hours for 3 days.
  Interventions: Drug: Rotigotine, Period 2

INTERVENTIONS:
Drug: Rotigotine, Period 1 — Formulation: transdermal
  Dosage: 2 mg / 24 hours once at Day 2
  Frequency: once every 24 hours
  Duration: from Day 1 to Day 3
  Other Names: Neupro
  Arms: Rotigotine, Period 1
Drug: Rotigotine, Period 2 — Formulation: transdermal
  Dosage: 2 mg / 24 hours for 3 days from Day 7 to Day 9, 4 mg / 24 hours for 3 days from Day 10 to Day 12
  Frequency: once every 24 hours
  Duration: from Day 1 to Day 3
  Other Names: Neupro
  Arms: Rotigotine, Period 2

SUMMARY:
This study is to characterize the Pharmacokinetics (PK) of unconjugated and total Rotigotine after single and multiple doses of Rotigotine transdermal patch, and also to investigate the safety and tolerability of Rotigotine transdermal patch in healthy Chinese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Chinese subjects
* Healthy volunteers with normal body weight, female subject is willing to use a double contraceptive barrier method or an oral hormonal contraceptive during the entire study

Exclusion Criteria:

* Previously participated in any Rotigotine study or participated in another clinical study for an investigational drug
* History of drug or alcohol abuse within the last 2 years
* Suicide attempt or suicidal ideation in the past 6 months
* Transient ischemic attack or stroke within the last 12 months
* Current condition of epilepsy and / or seizures
* History of significant skin hypersensitivity to adhesives or other transdermal products or recently unsolved contact dermatitis
* History or present condition of an atopic or eczematous dermatitis, psoriasis and / or an active skin disease
* Female subject is pregnant or lactating
* Subject has any medical or psychiatric condition that, in the opinion of the investigator, could jeopardize or would compromise the subject's wellbeing or ability to participate in this study
* Subject has a QTcB (QT interval corrected for heart rate according to Bazett's formula) interval of ≥ 450 ms for female or ≥ 430 ms for male
* Subject has a relevant hepatic dysfunction (total bilirubin > 2 mg / dL or alanine aminotransferase [ALT] or aspartate aminotransferase [AST] greater than 2 times the upper limit of the normal reference range)
* Subject has tested positive for human immunodeficiency virus antibodies (HIV)-1 / 2Ab, hepatitis B surface antigen (HBsAg) or hepatitis C virus antibody (HCV-Ab)
* Subject has a positive urine drug screen and / or alcohol breath test on Day 1
* Subject has made a blood donation or had a comparable blood loss (> 400 mL)
* Subject smokes or has done so within 6 months prior to Eligibility Assessment (EA)
* Subject has a clinically relevant allergy
* Subject is currently taking any medication
* Female subject is currently taking an oral hormonal contraceptive
* Subject has symptomatic orthostatic hypotension
* Subject has a pulse rate at rest less than 45 beats per minute (bpm) or more than 100 bpm
* Subject has a systolic blood pressure (SBP) lower than 100 mmHg or higher than 140 mmHg or diastolic blood pressure (DBP) higher than 90 mmHg
* Subject has a current or a history of clinically relevant motor disturbance, impairment of memory, sleep disturbance or neurodegenerative disease
* Subject has consumed more than 3 cups (more than 450 ml) of caffeinated beverages per day
* Subject's abdomen is thickly covered with hair resulting in difficulties in finding appropriate patch application sites

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-08; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of unconjugated Rotigotine for single-dose application (Period 1) | Period 1; Day 1 to Day 3 of study
  Period 1; Pharmacokinetic (PK) samples will be taken predose and 1, 2, 3, 4, 8, 12, 16, 24, 25, 26, 28, 30, 32, 36, 40, 48, 60 and 72 hours after patch application on Day 1
Plasma concentrations of unconjugated Rotigotine for multiple-dose application (Period 2) | Period 2; Day 7 to Day 14 of study
  Period 2; Pharmacokinetic (PK) samples will be taken prior to patch application on Day 7, 8, 9, 11 and 12 and 1, 2, 3, 4, 8, 12, 16 and 24 hours after patch application on Day 9 and 12 and 25, 26, 28, 30, 32, 36, 40, 48, 60 and 72 hours after patch application on Day 12
Plasma concentrations of total Rotigotine for single-dose application (Period 1) | Period 1; Day 1 to Day 3 of study
  Period 1; Pharmacokinetic (PK) samples will be taken predose and 1, 2, 3, 4, 8, 12, 16, 24, 25, 26, 28, 30, 32, 36, 40, 48, 60 and 72 hours after patch application on Day 1
Plasma concentrations of total Rotigotine for multiple-dose application (Period 2) | Period 2; Day 7 to Day 14 of study
  Period 2; Pharmacokinetic (PK) samples will be taken prior to patch application on Day 7, 8, 9, 11 and 12 and 1, 2, 3, 4, 8, 12, 16 and 24 hours after patch application on Day 9 and 12 and 25, 26, 28, 30, 32, 36, 40, 48, 60 and 72 hours after patch application on Day 12
Area under the plasma concentration-time curve from zero up to the last analytically quantifiable concentration (AUC 0-tz) for single-dose application (Period 1) | Period 1; Day 1 to Day 3 of study
  Period 1; Pharmacokinetic (PK) samples will be taken predose and 1, 2, 3, 4, 8, 12, 16, 24, 25, 26, 28, 30, 32, 36, 40, 48, 60 and 72 hours after patch application on Day 1
Maximum plasma concentration (Cmax) for single-dose application (Period 1) | Period 1; Day 1 to Day 3 of study
  Period 1; Pharmacokinetic (PK) samples will be taken predose and 1, 2, 3, 4, 8, 12, 16, 24, 25, 26, 28, 30, 32, 36, 40, 48, 60 and 72 hours after patch application on Day 1
Area under the plasma concentration-time curve from zero to 24 hours at steady state (AUC(0-24h),ss) for multiple-dose application (Period 2) | Period 2; Day 9 to Day 12 of study for this Primary Outcome Measure
  Period 2; Pharmacokinetic (PK) samples will be taken prior to patch application and 1, 2, 3, 4, 8, 12, 16 and 24 hours after patch application on Day 9 and Day 12
Maximum plasma concentration at steady state (Cmax,ss) for multiple-dose application (Period 2) | Period 2; Day 9 to Day 12 of study for this Primary Outcome Measure
  Period 2; Pharmacokinetic (PK) samples will be taken prior to patch application and 1, 2, 3, 4, 8, 12, 16 and 24 hours after patch application on Day 9 and Day 12

SECONDARY OUTCOMES:
Terminal half-life (t½) for single-dose application (Period 1) | Period 1; Day 1 to Day 3 of study
  Period 1; Pharmacokinetic (PK) samples will be taken predose and 1, 2, 3, 4, 8, 12, 16, 24, 25, 26, 28, 30, 32, 36, 40, 48, 60 and 72 hours after patch application on Day 1
Time to reach a maximum plasma concentration (tmax) for single-dose application (Period 1) | Period 1; Day1 to Day 3 of study
  Period 1; Pharmacokinetic (PK) samples will be taken predose and 1, 2, 3, 4, 8, 12, 16, 24, 25, 26, 28, 30, 32, 36, 40, 48, 60 and 72 hours after patch application on Day 1
Lag time until first concentration ≥ limit of quantitation (LOQ) (tlag) for single-dose application (Period 1) | Period 1; Day 1 to Day 3 of study
  Period 1; Pharmacokinetic (PK) samples will be taken predose and 1, 2, 3, 4, 8, 12, 16, 24, 25, 26, 28, 30, 32, 36, 40, 48, 60 and 72 hours after patch application on Day 1
Maximum plasma concentration normalized by Body Weight (kg) (Cmax, norm (BW)) for single-dose application (Period 1) | Period 1; Day 1 to Day 3 of study
  Period 1; Pharmacokinetic (PK) samples will be taken predose and 1, 2, 3, 4, 8, 12, 16, 24, 25, 26, 28, 30, 32, 36, 40, 48, 60 and 72 hours after patch application on Day 1
Maximum plasma concentration normalized by apparent dose (mg)(Cmax, norm (apparent dose)) for single-dose application (Period 1) | Period 1; Day 1 to Day 3 of study
  Period 1; Pharmacokinetic (PK) samples will be taken predose and 1, 2, 3, 4, 8, 12, 16, 24, 25, 26, 28, 30, 32, 36, 40, 48, 60 and 72 hours after patch application on Day 1
Maximum plasma concentration normalized by drug content of patch (mg) (Cmax, norm (mgdc)) for single-dose application (Period 1) | Period 1; Day 1 to Day 3 of study
  Period 1; Pharmacokinetic (PK) samples will be taken predose and 1, 2, 3, 4, 8, 12, 16, 24, 25, 26, 28, 30, 32, 36, 40, 48, 60 and 72 hours after patch application on Day 1
Area under the plasma concentration-time curve from zero up to the last analytically quantifiable concentration normalized by body weight (kg) (AUC(0-tz), norm (BW)) for single-dose application (Period 1) | Perion 1; Day 1 to Day 3 of study
  Period 1; Pharmacokinetic (PK) samples will be taken predose and 1, 2, 3, 4, 8, 12, 16, 24, 25, 26, 28, 30, 32, 36, 40, 48, 60 and 72 hours after patch application on Day 1
Area under the plasma concentration-time curve from zero up to the last analytically quantifiable concentration normalized by apparent dose (mg) (AUC(0-tz), norm (apparent dose)) for single-dose application (Period 1) | Period 1; Day 1 to Day 3 of study
  Period 1; Pharmacokinetic (PK) samples will be taken predose and 1, 2, 3, 4, 8, 12, 16, 24, 25, 26, 28, 30, 32, 36, 40, 48, 60 and 72 hours after patch application on Day 1
Area under the plasma concentration-time curve from zero up to the last analytically quantifiable concentration normalized by drug content of patch (mg) (AUC(0-tz), norm (mgdc)) for single-dose application (Period 1) | Period 1; Day 1 to Day 3 of study
  Period 1; Pharmacokinetic (PK) samples will be taken predose and 1, 2, 3, 4, 8, 12, 16, 24, 25, 26, 28, 30, 32, 36, 40, 48, 60 and 72 hours after patch application on Day 1
Area under the plasma concentration-time curve from zero up to infinity (AUC(0-∞)) for single-dose application (Period 1) | Period 1; Day 1 to Day 3 of study
  Period 1; Pharmacokinetic (PK) samples will be taken predose and 1, 2, 3, 4, 8, 12, 16, 24, 25, 26, 28, 30, 32, 36, 40, 48, 60 and 72 hours after patch application on Day 1
Area under the plasma concentration-time curve from zero up to infinity normalized by apparent dose (mg) (AUC(0-∞), norm (apparent dose)) for single-dose application (Period 1) | Period 1; Day 1 to Day 3 of study
  Period 1; Pharmacokinetic (PK) samples will be taken predose and 1, 2, 3, 4, 8, 12, 16, 24, 25, 26, 28, 30, 32, 36, 40, 48, 60 and 72 hours after patch application on Day 1
Area under the plasma concentration-time curve from zero up to infinity normalized by body weight (kg) (AUC(0-∞), norm (BW)) for single-dose application (Period 1) | Period 1; Day 1 to Day 3 of study
  Period 1; Pharmacokinetic (PK) samples will be taken predose and 1, 2, 3, 4, 8, 12, 16, 24, 25, 26, 28, 30, 32, 36, 40, 48, 60 and 72 hours after patch application on Day 1
Area under the plasma concentration-time curve from zero up to infinity normalized by drug content of patch (mg) (AUC(0-∞), norm (mgdc)) for single-dose application (Period 1) | Period 1; Day 1 to Day 3 of study
  Period 1; Pharmacokinetic (PK) samples will be taken predose and 1, 2, 3, 4, 8, 12, 16, 24, 25, 26, 28, 30, 32, 36, 40, 48, 60 and 72 hours after patch application on Day 1
Apparent total body clearance (CL/F) for single-dose application (Period 1) | Period 1; Day 1 to Day 3 of study
  Period 1; Pharmacokinetic (PK) samples will be taken predose and 1, 2, 3, 4, 8, 12, 16, 24, 25, 26, 28, 30, 32, 36, 40, 48, 60 and 72 hours after patch application on Day 1
Apparent total body clearance normalized by body weight (kg) (CL/F norm (BW)) for single-dose application (Period 1) | Period 1; Day 1 to Day 3 of study
  Period 1; Pharmacokinetic (PK) samples will be taken predose and 1, 2, 3, 4, 8, 12, 16, 24, 25, 26, 28, 30, 32, 36, 40, 48, 60 and 72 hours after patch application on Day 1
Apparent volume of distribution (Vz/f) for single-dose application (Period 1) | Period 1; Day 1 to Day 3 of study
  Period 1; Pharmacokinetic (PK) samples will be taken predose and 1, 2, 3, 4, 8, 12, 16, 24, 25, 26, 28, 30, 32, 36, 40, 48, 60 and 72 hours after patch application on Day 1
Apparent volume of distribution normalized by body weight (kg) (Vz/f norm (BW)) for single-dose application (Period 1) | Period 1; Day 1 to Day 3 of study
  Period 1; Pharmacokinetic (PK) samples will be taken predose and 1, 2, 3, 4, 8, 12, 16, 24, 25, 26, 28, 30, 32, 36, 40, 48, 60 and 72 hours after patch application on Day 1
Mean residence time (MRT) for single-dose application (Period 1) | Period 1; Day 1 to Day 3 of study
  Period 1; Pharmacokinetic (PK) samples will be taken predose and 1, 2, 3, 4, 8, 12, 16, 24, 25, 26, 28, 30, 32, 36, 40, 48, 60 and 72 hours after patch application on Day 1
Rate constant of elimination (ke) for single-dose application (Period 1) | Period 1; Day 1 to Day 3 of study
  Period 1; Pharmacokinetic (PK) samples will be taken predose and 1, 2, 3, 4, 8, 12, 16, 24, 25, 26, 28, 30, 32, 36, 40, 48, 60 and 72 hours after patch application on Day 1
Terminal half-life (t½) for multiple-dose application | Period 2; Day 7 to Day 14 of study
  Period 2; Pharmacokinetic (PK) samples will be taken prior to patch application on Day 7, 8, 9, 11 and 12 and 1, 2, 3, 4, 8, 12, 16 and 24 hours after patch application on Day 9 and 12 and 25, 26, 28, 30, 32, 36, 40, 48, 60 and 72 hours after patch application on Day 12
Time to reach a maximum plasma concentration at steady state (tmax,ss) for multiple-dose application (Period 2) | Period 2; Day 9 to Day 12 of study for this Outcome Measure.
  Period 2; Pharmacokinetic (PK) samples will be taken prior to patch application on Day 9 and Day 12 and 1, 2, 3, 4, 8, 12, 16 and 24 hours after patch application on Day 9 and Day 12
Maximum plasma concentration at steady state normalized by body weight (kg) (Cmax,ss,norm(BW)) for multiple-dose application (Period 2) | Period 2; Day 9 to Day 12 of study for this Outcome Measure.
  Period 2; Pharmacokinetic (PK) samples will be taken prior to patch application on Day 9 and Day 12 and 1, 2, 3, 4, 8, 12, 16 and 24 hours after patch application on Day 9 and Day 12
Maximum plasma concentration at steady state normalized by apparent dose (mg) (Cmax, ss, norm (apparent dose)) for multiple-dose application (Period 2) | Period 2; Day 9 to Day 12 of study for this Outcome Measure.
  Period 2; Pharmacokinetic (PK) samples will be taken prior to patch application on Day 9 and Day 12 and 1, 2, 3, 4, 8, 12, 16 and 24 hours after patch application on Day 9 and Day 12
Maximum plasma concentration at steady state normalized by drug content of patch (mg) (Cmax, ss, norm (mgdc)) for multiple-dose application (Period 2) | Period 2; Day 9 to Day 12 of study for this Outcome Measure
  Period 2; Pharmacokinetic (PK) samples will be taken prior to patch application on Day 9 and Day 12 and 1, 2, 3, 4, 8, 12, 16 and 24 hours after patch application on Day 9 and Day 12
Minimum plasma concentration at steady state (Cmin, ss) for multiple-dose application (Period 2) | Period 2; Day 9 to Day 12 of study for this Outcome Measure
  Period 2; Pharmacokinetic (PK) samples will be taken prior to patch application on Day 9 and Day 12 and 1, 2, 3, 4, 8, 12, 16 and 24 hours after patch application on Day 9 and Day 12
Area under the plasma concentration-time curve from zero to 24 hours at steady state normalized by body weight (kg) (AUC(0-24h), ss, norm (BW)) for multiple-dose application (Period 2) | Period 2; Day 9 to Day 12 of study for this Outcome Measure
  Period 2; Pharmacokinetic (PK) samples will be taken prior to patch application on Day 9 and Day 12 and 1, 2, 3, 4, 8, 12, 16 and 24 hours after patch application on Day 9 and Day 12
Area under the plasma concentration-time curve from zero to 24 hours at steady state normalized by apparent dose (mg) (AUC(0-24), ss, norm (apparent dose)) for multiple-dose application (Period 2) | Period 2; Day 9 to Day 12 of study for this Outcome Measure
  Period 2; Pharmacokinetic (PK) samples will be taken prior to patch application on Day 9 and Day 12 and 1, 2, 3, 4, 8, 12, 16 and 24 hours after patch application on Day 9 and Day 12
Area under the plasma concentration-time curve from zero to 24 hours at steady state normalized by drug content of patch (mg) (AUC(0-24), ss, norm (mgdc)) for multiple-dose application (Period 2) | Period 2; Day 9 to Day 12 of study for this Outcome Measure
  Period 2; Pharmacokinetic (PK) samples will be taken prior to patch application on Day 9 and Day 12 and 1, 2, 3, 4, 8, 12, 16 and 24 hours after patch application on Day 9 and Day 12
Apparent total body clearance (CL/F) for multiple-dose application (Period 2) | Period 2; Day 7 to Day 14 of study
  Period 2; Pharmacokinetic (PK) samples will be taken prior to patch application on Day 7, 8, 9, 11 and 12 and 1, 2, 3, 4, 8, 12, 16 and 24 hours after patch application on Day 9 and Day 12 and 25, 26, 28, 30, 32, 36, 40, 48, 60 and 72 hours on Day 12.
Apparent total body clearance normalized by body weight (kg) (CL/F norm (BW)) for multiple-dose application (Period 2) | Period 2; Day 7 to Day 14 of study
  Period 2; Pharmacokinetic (PK) samples will be taken prior to patch application on Day 7, 8, 9, 11 and 12 and 1, 2, 3, 4, 8, 12, 16 and 24 hours after patch application on Day 9 and Day 12 and 25, 26, 28, 30, 32, 36, 40, 48, 60 and 72 hours on Day 12.
Apparent volume of distribution (Vz/f) for multiple-dose application (Period 2) | Period 2; Day 7 to Day 14 of study
  Period 2; Pharmacokinetic (PK) samples will be taken prior to patch application on Day 7, 8, 9, 11 and 12 and 1, 2, 3, 4, 8, 12, 16 and 24 hours after patch application on Day 9 and Day 12 and 25, 26, 28, 30, 32, 36, 40, 48, 60 and 72 hours on Day 12.
Apparent volume of distribution normalized by body weight (kg) (Vz/f norm (BW)) for multiple-dose application (Period 2) | Period 2; Day 7 to Day 14 of study
  Period 2; Pharmacokinetic (PK) samples will be taken prior to patch application on Day 7, 8, 9, 11 and 12 and 1, 2, 3, 4, 8, 12, 16 and 24 hours after patch application on Day 9 and Day 12 and 25, 26, 28, 30, 32, 36, 40, 48, 60 and 72 hours on Day 12.
Mean residence time (MRT) for multiple-dose application (Period 2) | Period 2; Day 7 to Day 14 of study
  Period 2; Pharmacokinetic (PK) samples will be taken prior to patch application on Day 7, 8, 9, 11 and 12 and 1, 2, 3, 4, 8, 12, 16 and 24 hours after patch application on Day 9 and Day 12 and 25, 26, 28, 30, 32, 36, 40, 48, 60 and 72 hours on Day 12.
Rate constant of elimination (ke) for multiple-dose application (Period 2) | Period 2; Day 7 to Day 14 of study
  Period 2; Pharmacokinetic (PK) samples will be taken prior to patch application on Day 7, 8, 9, 11 and 12 and 1, 2, 3, 4, 8, 12, 16 and 24 hours after patch application on Day 9 and Day 12 and 25, 26, 28, 30, 32, 36, 40, 48, 60 and 72 hours on Day 12.
Peak to trough fluctuation (PTF) for multiple-dose application (Period 2) | Period 2; Day 9 to Day 12 of study for this Outcome Measure
  Period 2; Pharmacokinetic (PK) samples will be taken prior to patch application on Day 9 and Day 12 and 1, 2, 3, 4, 8, 12, 16 and 24 hours after patch application on Day 9 and Day 12.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai, China

REFERENCES:
- [Derived] Liu Y, Tomlinson B, Guo J, Asgharnejad M, Bauer L, Surmann E, Guo X, Elshoff JP. Pharmacokinetics, Tolerability, and Bioequivalence of Two Formulations of Rotigotine in Healthy Chinese Subjects. Clin Ther. 2018 Jul;40(7):1108-1121.e8. doi: 10.1016/j.clinthera.2018.05.009. PMID 30098648